CLINICAL TRIAL: NCT03797781
Title: Understanding the Role of Protein Ingestion on Skeletal Muscle Atrophy During an Acute Period of Disuse
Brief Title: Protein Ingestion and Skeletal Muscle Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 6500619582
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High protein (Experimental)
  Interventions: Other: Lower limb immobilisation (leg brace) with varying levels of protein intake
- Low protein (Experimental)
  Interventions: Other: Lower limb immobilisation (leg brace) with varying levels of protein intake
- Minimum protein (Experimental)
  Interventions: Other: Lower limb immobilisation (leg brace) with varying levels of protein intake

INTERVENTIONS:
Other: Lower limb immobilisation (leg brace) with varying levels of protein intake — Single leg immobilisation via leg brace and crutches, the groups have different amounts of protein intake

SUMMARY:
The effect of different protein intakes on skeletal muscle atrophy during short term unilateral leg immobilisation.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18 and <28 no prescription medications or current illness.

Exclusion Criteria:

* BMI <18 and >28 current prescription medication no history of leg injury.
* Smoker
* Medical conditions including (cardiovascular disease ((e.g. hypertension)), metabolic disease ((e.g. type 2 diabetes)), any personal or family history of deep vein thrombosis.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle size | 3 days

SECONDARY OUTCOMES:
Muscle strength | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Health Science, Exeter, Devon, United Kingdom

REFERENCES:
- [Derived] Kilroe SP, Fulford J, Jackman S, Holwerda A, Gijsen A, van Loon L, Wall BT. Dietary protein intake does not modulate daily myofibrillar protein synthesis rates or loss of muscle mass and function during short-term immobilization in young men: a randomized controlled trial. Am J Clin Nutr. 2021 Mar 11;113(3):548-561. doi: 10.1093/ajcn/nqaa136. PMID 32469388